CLINICAL TRIAL: NCT06342128
Title: Comprehensive Multiscale Characterization of the Molecular Landscape of Microvascular Inflammation in Kidney Allografts
Brief Title: Molecular Landscape of Microvascular Inflammation in Kidney Allografts
Status: Recruiting | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: MVI_Kidney_001
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2024-11

CONDITIONS: Kidney Rejection Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Microvascular inflammation in kidney allografts has been widely reappraised in the recent update of Banff classification. There is a critical need to better understand the pathophysiological mechanisms associated with the various phenotypes of microvascular inflammation that are observed in kidney transplants, particularly in order to develop targeted therapeutic approaches.

DETAILED DESCRIPTION:
Antibody-mediated rejection is a major cause of graft failure in kidney transplant recipients. The diagnostic criteria for antibody-mediated rejection have undergone significant changes since their initial definition in the international Banff Classification system. The Banff 2022 Classification update reappraises lesions of microvascular inflammation and identifies new phenotypes for cases with microvascular inflammation. However, pathophysiological mechanisms associated with microvascular inflammation in kidney allografts are still poorly understood, thus hampering the development of efficient treatments.

The aims of this study are:

1. To decipher the spatial immune-molecular landscape of microvascular inflammation in kidney allografts.
2. To compare the characteristics of this landscape in different clinical scenarios.

The investigators will use a multimodal phenotyping approach including histological analyses and multiplex immunostainings, bulk transcriptomic analyses and spatial whole-transcriptome digital profiling to decipher the molecular landscape of microvascular inflammation in kidney allografts. Based on these results, they will investigate its association with allograft outcomes and search for molecular targets which could benefit from targeted therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

- Adult kidney transplant recipients, with at least one kidney transplant biopsy performed and assessed according to the international Banff 2022 classification, with or without lesions of microvascular inflammation

Exclusion Criteria:

* Inadequate biopsy according to the Banff classification
* Missing data for Banff lesion scores, donor-specific antibody status, C4d staining
* Biopsies showing histological signs of ischemia-reperfusion
* Combined transplantation and kidney transplantation after a non-kidney solid organ transplantation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult kidney transplant recipients of all sexes (self-determined) recruited in Europe and United States, who had a kidney allograft biopsy with or without lesions of microvascular inflammation (adequate biopsies without missing data for Banff lesion scores, donor-specific antibody status, and C4d staining), according to the international Banff 2022 classification.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
RNA-based molecular signatures assessed using bulk and spatial transcriptomics | 1 day (at time of a kidney allograft biopsy)
Probability of graft survival based on outcome data | 24 months post-kidney allograft biopsy
Probability of patient survival on outcome data | 24 months post-kidney allograft biopsy

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Kidney Transplant Department, Saint-Louis Hospital, Assistance Publique - Hôpitaux de Paris, Paris
  - Kidney Transplant Department, Necker Hospital, Assistance Publique - Hôpitaux de Paris, Paris
  - Bichat Hospital, Assistance Publique - Hôpitaux de Paris, Paris

IPD SHARING:
Plan to Share IPD: Undecided
The data analyzed during the current study are available on reasonable request including standards for General Data Protection Regulation and Institutional Review Board approval.

REFERENCES:
- [Background] Loupy A, Haas M, Roufosse C, Naesens M, Adam B, Afrouzian M, Akalin E, Alachkar N, Bagnasco S, Becker JU, Cornell LD, Clahsen-van Groningen MC, Demetris AJ, Dragun D, Duong van Huyen JP, Farris AB, Fogo AB, Gibson IW, Glotz D, Gueguen J, Kikic Z, Kozakowski N, Kraus E, Lefaucheur C, Liapis H, Mannon RB, Montgomery RA, Nankivell BJ, Nickeleit V, Nickerson P, Rabant M, Racusen L, Randhawa P, Robin B, Rosales IA, Sapir-Pichhadze R, Schinstock CA, Seron D, Singh HK, Smith RN, Stegall MD, Zeevi A, Solez K, Colvin RB, Mengel M. The Banff 2019 Kidney Meeting Report (I): Updates on and clarification of criteria for T cell- and antibody-mediated rejection. Am J Transplant. 2020 Sep;20(9):2318-2331. doi: 10.1111/ajt.15898. Epub 2020 May 28. PMID 32463180
- [Background] Mengel M, Loupy A, Haas M, Roufosse C, Naesens M, Akalin E, Clahsen-van Groningen MC, Dagobert J, Demetris AJ, Duong van Huyen JP, Gueguen J, Issa F, Robin B, Rosales I, Von der Thusen JH, Sanchez-Fueyo A, Smith RN, Wood K, Adam B, Colvin RB. Banff 2019 Meeting Report: Molecular diagnostics in solid organ transplantation-Consensus for the Banff Human Organ Transplant (B-HOT) gene panel and open source multicenter validation. Am J Transplant. 2020 Sep;20(9):2305-2317. doi: 10.1111/ajt.16059. Epub 2020 Jun 27. PMID 32428337
- [Background] Loupy A, Mengel M, Haas M. Thirty years of the International Banff Classification for Allograft Pathology: the past, present, and future of kidney transplant diagnostics. Kidney Int. 2022 Apr;101(4):678-691. doi: 10.1016/j.kint.2021.11.028. Epub 2021 Dec 17. PMID 34922989
- [Background] Naesens M, Roufosse C, Haas M, Lefaucheur C, Mannon RB, Adam BA, Aubert O, Bohmig GA, Callemeyn J, Clahsen-van Groningen M, Cornell LD, Demetris AJ, Drachenberg CB, Einecke G, Fogo AB, Gibson IW, Halloran P, Hidalgo LG, Horsfield C, Huang E, Kikic Z, Kozakowski N, Nankivell B, Rabant M, Randhawa P, Riella LV, Sapir-Pichhadze R, Schinstock C, Solez K, Tambur AR, Thaunat O, Wiebe C, Zielinski D, Colvin R, Loupy A, Mengel M. The Banff 2022 Kidney Meeting Report: Reappraisal of microvascular inflammation and the role of biopsy-based transcript diagnostics. Am J Transplant. 2024 Mar;24(3):338-349. doi: 10.1016/j.ajt.2023.10.016. Epub 2023 Oct 28. PMID 38032300